CLINICAL TRIAL: NCT00407121
Title: Intravitreal Bevacizumab for the Treatment of Neovascular Membranes in Patients With Intraocular Inflammation
Brief Title: Intravitreal Bevacizumab for Inflammatory Neovascular Membranes
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Undefined.
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APEC-0025
Record Dates: First submitted 2006-12-01; First posted 2006-12-04 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Vogt Koyanagi Harada Disease; Serpiginous Choroiditis; Multifocal Choroiditis
Keywords: Neovascular Membrane; Uveitis; Bevacizumab
MeSH Terms: conditions — Uveomeningoencephalitic Syndrome; White Dot Syndromes; Multifocal Choroiditis; Uveitis | interventions — Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab
Procedure: Intravitreal Injection of Bevacizumab

SUMMARY:
Intravitreal injection of Bevacizumab in patients with Neovascular Membranes secondary to intraocular inflammation. We injected a single injection of Bevacizumab (2.5 mg/0.1 ml) and evaluate visual acuity , Fluorescein angiogram and retinal thickness by Optical Coherence Tomography (OCT) in 4 patients with Vogt Koyanagi Harada disease, 1 patient with Serpiginous Choroidopathy and 1 patient with Multifocal Choroiditis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnose
* Patient Consent
* Chronic stage of inflammation

Exclusion Criteria:

* only eye
* age lower than 30 yo.
* Systemic condition

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-12 (Actual); Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity
Retinal thickness by OCT
Leakage in Fluorescein angiogram

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Kon-Jara, MD, Principal Investigator — Asociación para Evitar la Ceguera en México; LuzElena Concha-Del Rio, MD, Study Chair — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociacion para Evitar la Ceguera en Mexico, Mexico City, Mexico City, Mexico